CLINICAL TRIAL: NCT06247930
Title: Effect of Vitamin D Supplementation on Depressive Symptoms in Chinese Early Adolescents
Brief Title: An Evaluation of the Effect of Vitamin D Supplementation on Depressive Symptoms Among Chinese Early Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yuan Mengyuan, Principal Investigator, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 84230079
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-09

CONDITIONS: Depressive Symptoms
Keywords: depressive symptoms; vitamin D
MeSH Terms: conditions — Depression | interventions — Cholecalciferol; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 + Mental Health Education (Experimental): Vitamin D3: 2000 IU per day for 6 weeks (two capsules of 800 IU plus one capsule of 400 IU), followed by 800 IU (one capsule of 800 IU) per day for 6 weeks.
  Mental Health Education: consists of providing a brochure and videos containing information about mental health problems.
  Interventions: Dietary Supplement: Vitamin D3; Behavioral: Mental health education
- Vitamin D3 placebo + Mental Health Education (Placebo Comparator): Vitamin D3 placebo (i.e., soybean oil). Mental Health Education: consists of providing a brochure and videos containing information about mental health problems.
  Interventions: Dietary Supplement: Vitamin D3 placebo; Behavioral: Mental health education

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 2000 IU per day for 6 weeks (two capsules of 800 IU plus one capsule of 400 IU), followed by 800 IU (one capsule of 800 IU) per day for 6 weeks.
  Other Names: Cholecalciferol
  Arms: Vitamin D3 + Mental Health Education
Dietary Supplement: Vitamin D3 placebo — Three capsules for 6 weeks, followed by one capsule for 6 weeks.
  Other Names: Soybean oil
  Arms: Vitamin D3 placebo + Mental Health Education
Behavioral: Mental health education — The mental health education consists of providing a brochure and videos containing information about mental health problems.

SUMMARY:
The goal of this randomized controlled clinical trial is to investigate the effects of vitamin D3 supplementation on depression in Chinese early adolescents with elevated depressive symptoms and vitamin D deficiency. The main question it aims to answer whether vitamin D3 supplementation can reduce depressive symptoms.

Participants in the intervention group will receive vitamin D3 capsules and mental health education. The control group will receive vitamin D3 placebo and mental health education.

Researchers will compare the change in depressive symptoms from baseline to post-intervention at 12 weeks between the intervention and control groups.

DETAILED DESCRIPTION:
Investigators will conduct a randomized controlled trial to examine whether vitamin D3 supplementation can improve depressive symptoms. Participants will be recruited from two middle schools. Participants will be randomly assigned into a supplementation or placebo group. Supplementation arm will receive oral dose 2000 IU vitamin D3 per day for 6 weeks and followed by 800 IU per day for 6 weeks; placebo arm will receive placebo every day for 12 weeks. Both of these two groups will receive additional mental health education. For the first 6 weeks, vitamin D or placebo will be administrated every two weeks. For the next 6 weeks, vitamin D or placebo will be administrated every three weeks. The primary outcome of this study is to compare the change of depressive symptoms between supplementation or placebo group from pre- to post-intervention at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 7th-9th students whose caregivers signed informed consents;
2. students with serum 25(OH)D concentrations below 20 ng/mL;
3. students with self-reported depressive symptoms (BDI-II score of 14 or higher)

Exclusion Criteria:

1. students who are currently receiving or have used anti-psychotic treatments or interventions (including drugs and non-drugs) in the past 3 months;
2. students who have serious health conditions (e.g., organic or functional brain diseases, major psychiatric disorders, cardiovascular diseases, serious infectious diseases, chronic gastrointestinal diseases, and hepatic or renal diseases);
3. students who are currently taking or have taken vitamin D supplements in the past 3 months;
4. students with self-reported serious suicidal ideation, suicidal plans and attempts in the past 3 months;
5. students with intellectual disability;
6. students who are allergic to vitamin D or soybean oil components.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 406 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptom scores | From randomization to the end of intervention at 3 months
  Depressive symptoms are evaluated by the Chinese version of Beck Depression Inventory (BDI-II-C). The measured outcome was the total BDI-II-C scores. Each of the 21 items can be scored as 0, 1, 2, or 3 points. The range for the BDI-II-C score is 0-63 points; higher scores indicate worse depressive symptoms. Change in BDI-II-C scores from pre to post-intervention were compared between randomized groups, which was the primary outcome of this study.

SECONDARY OUTCOMES:
Depressive Symptoms Scores | Baseline, 6, 9, 24 and 36 weeks
  Depressive symptoms are assessed by BDI-II-C. Data from all time points will be used to determine the mean differences in change in depressive symptoms scores over all follow-up by randomized treatment.
Patient Health Questionnaire-9 Scores | Baseline, 6, 9, 12, 24 and 36 weeks
  Patient Health Questionnaire-9 (PHQ-9) is a 9-item instrument for measuring the severity of depression. The PHQ-9 is based on the diagnosis of the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) depressive disorders. Each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day), and the total scores of PHQ-9 can range from 0 to 27. The higher score indicates more depressive symptoms. It can be administrated repeatedly and can reflect improvement or worsening of depression in response to treatment. Data from all time points will be used to determine the mean differences in change in depression scores over all follow-up by randomized treatment.
Sleep Quality Scores | Baseline, 6, 12, 24 and 36 weeks
  Sleep quality is evaluated by the Pittsburgh Sleep Quality Index (PSQI). In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality. Data from all time points will be used to determine the mean differences in change in sleep quality scores over all follow-up by randomized treatment.
Number of Participants with a Suicidal Ideation Event | From randomization to the occurrence of the endpoint or to the end of evaluation at 12, 24 or 36 weeks.
  Suicidal ideation will be asked by the item 'In the past three months, have you ever thought about killing yourself?'. The responses will be classified as yes or no.
Anxiety Symptoms Scores | Baseline, 6, 9, 12, 24 and 36 weeks
  Anxiety symptoms will be assessed by the Generalized Anxiety Disorder 7-item scale (GAD-7). GAD-7 has seven items and assess the severity of the severity of generalized anxiety symptoms over the past two weeks. Response options include "not at all", "several days", "more than half the days" and "nearly every day". In scoring the GAD-7, each of seven items scored 0 (not at all), 1 (several days), 2 (more than half the days), and 3 (nearly every day). The total scores are calculated and range from 0 to 21. Higher scores indicate worse anxiety symptoms. Data from all time points will be used to determine the mean differences in change in sleep quality scores over all follow-up by randomized treatment.
Psychological Resilience Scores | Baseline, 6, 12 weeks
  Resilience will be evaluated by the Connor-Davidson Resilience Scale (CD-RISC). The CD-RISC consists of 25 items, which are evaluated on a five-point Likert scale ranging from 0 to 4: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4) - these ratings result in a number between 0-100, and higher scores indicate higher resilience. Data from all time points will be used to determine the mean differences in change in resilience scores over all follow-up by randomized treatment.
Hopelessness Scores | Baseline, 6, 12, 24 and 36 weeks
  Hopelessness will be evaluated by the Beck Hopelessness Scale (BHS). The BHS consists of 20 dichotomous "true/false" items that aims to assess three major aspects of hopelessness (i.e., feelings about the future, loss of motivation, and expectations). Higher total scores indicate greater hopelessness (range 0-20). Data from all time points will be used to determine the mean differences in change in hopelessness scores over all follow-up by randomized treatment.
Emotional and Behavioral Problems Scores | Baseline, 6, 9, 12, 24, 36 weeks
  Emotional and behavioral problems are assessed by the Pediatric Symptom Checklist-17 (PSC-17). The PSC-17 consists of 17 items, and is categorized as three subscales (5 items on internalizing subscale, 5 items on attention subscale, and 7 items on externalizing subscale). The responses are 0 ("Never"), 1 ("Sometimes") and 2 ("Often"). The total score of the PSC-17 is calculated, and ranges from 0 to 34. Higher scores can indicate an increased likelihood of a behavioral health disorder being present. Data from all time points will be used to determine the mean differences in change in internalizing, attention and externalizing scores over all follow-up by randomized treatment.
Loneliness Scores | Baseline, 6, 12, 24, 36 weeks
  Loneliness will be measured by the short-form University of California, Los Angeles (UCLA) Loneliness Scale (ULS-8). The total score ranges from 8 to 32 points, with higher scores suggesting a higher degree of loneliness. Data from all time points will be used to determine the mean differences in change in loneliness scores over all follow-up by randomized treatment.
Emotional Regulation Ability Scores | Baseline, 6, 12 weeks
  The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) is a 10-item scale to measure respondents' tendency to regulate their emotions and the total scores will be used in this study. Items are rated on a 5-point Likert-type response scale (1=strongly disagree, 2=disagree, 3=half and half, 4=agree and 5=strongly agree). The total score ranges from 10 to 50. Higher scores indicate greater use of the emotional regulation strategy. Data from all time points will be used to determine the mean differences in change in emotional regulation scores over all follow-up by randomized treatment.

OTHER OUTCOMES:
Irritability Scores | Baseline, 12, 36 weeks
  Irritability will be measured by the Affective Reactivity Index (ARI). The ARI scale contains six symptom items. Respondents rate irritability over the last 3 months. Each item has a three-level response category: 'not true', 'somewhat true', 'certainly true'- scored as '0', '1', '2', respectively, giving a range of possible scores of 0-12. The total scores will be calculated and used in this study. Data from all time points will be used to determine the mean differences in change in irritability scores over all follow-up by randomized treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Puyu Su, Professor, Principal Investigator — Anhui Medical University
Locations (2):
- China (2):
  - Susong County Guangfu Middle School, Anqing, Anhui
  - Susong County Zhenxing School, Anqing, Anhui

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be only used in a peer-reviewed journal in order to protect the privacy of the study participants.